CLINICAL TRIAL: NCT02504827
Title: Steady-state Pharmacokinetics of Ceftazidime/Avibactam in CF
Brief Title: Steady-state Pharmacokinetics of Ceftazidime/Avibactam in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Paul Beringer, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APP-15-01273
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
Keywords: pharmacokinetics; ceftazidime/avibactam
MeSH Terms: conditions — Cystic Fibrosis | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV Ceftazidime/Avibactam (Experimental): Ceftazidime/avibactam 2.5gm IV q8h for 3 doses
  Interventions: Drug: Ceftazidime/avibactam

INTERVENTIONS:
Drug: Ceftazidime/avibactam — Ceftazidime/avibactam 2.5gm iv q8h for 3 doses
  Other Names: Avycaz

SUMMARY:
The purpose of this research study is to characterize the pharmacokinetics of intravenous ceftazidime/avibactam in patients with Cystic Fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis is a genetic disorder characterized by a chronic cycle of airway infection, obstruction, and inflammation leading to progressive loss of lung function and eventual respiratory failure. The principal pathogen is Pseudomonas aeruginosa which is present in the airways of 70% of adult patients with CF. Of particular concern is the increasing resistance observed to existing agents.

While ceftazidime has been the mainstay of treatment for many years, its efficacy is limited by reduced susceptibility. Ceftazidime/avibactam offers a potential advancement in the management of infections involving P. aeruginosa in CF due to its excellent activity, penetration into pulmonary secretions, and reduced potential for development of resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on positive sweat chloride or know CF mutation
* Age > 17 years
* Able to spontaneously expectorate sputum

Exclusion Criteria:

* Any clinically significant laboratory abnormality
* Presence of an ongoing acute pulmonary exacerbation
* Pregnancy
* Serious past allergy to a beta-lactam antibiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beringer, PharmD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Bensman TJ, Wang J, Jayne J, Fukushima L, Rao AP, D'Argenio DZ, Beringer PM. Pharmacokinetic-Pharmacodynamic Target Attainment Analyses To Determine Optimal Dosing of Ceftazidime-Avibactam for the Treatment of Acute Pulmonary Exacerbations in Patients with Cystic Fibrosis. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00988-17. doi: 10.1128/AAC.00988-17. Print 2017 Oct. PMID 28784670

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Ceftazidime/Avibactam
Started | 12
Completed | 11
Not Completed | 1
Not completed — Could not produce sputum | 1

BASELINE CHARACTERISTICS:
Arm/Group | IV Ceftazidime/Avibactam
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax)
Time Frame: 8 hours
Measure: Mean (Full Range); unit: mg/L
Arm/Group | IV Ceftazidime/Avibactam
Number analyzed (Participants) | 12
mg/L | 85.87 [61.8 to 111.2]

2. Primary Outcome: Peak Sputum Concentration
Time Frame: 8 hours
Measure: Mean (Full Range); unit: mg/L
Arm/Group | IV Ceftazidime/Avibactam
Number analyzed (Participants) | 11
mg/L | 2.5 [0.6 to 9.4]

ADVERSE EVENTS:
Arm/Group | IV Ceftazidime/Avibactam
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No